CLINICAL TRIAL: NCT07105566
Title: Serum Triosephosphate Isomerase Level in Pateints With Rheumatoid Arthritis : Relation to Disease Activity and Structural Damage
Brief Title: Triosephosphate Isomerase Level in Relation to Rheumatoid Aerthritis Activity and Structural Damage
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Mohsen Obeid Hassan, Principal Investigator, Assiut University
Other Study IDs: TPI level in RA patients
Record Dates: First submitted 2025-07-16; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- cases: Rheumatoid Arthritis pateints
  Interventions: Diagnostic Test: serum TPI
- controls: healthy controls
  Interventions: Diagnostic Test: serum TPI

INTERVENTIONS:
Diagnostic Test: serum TPI — serum TPI level
  Other Names: ultrasound

SUMMARY:
1. Assess the serum level of TPI in patients with RA compared to healthy controls.
2. Correlate serum level of TPI and disease activity.
3. Correlation of serum TPI level with US7 damage index

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic systemic autoimmune disease characterized by persistent synovial inflammation, synovial hyperplasia, and progressive destruction of bone and cartilage. These pathological processes can lead to joint deformities and loss of function, significantly affecting patients' quality of life. In addition to joint damage, RA often manifests with extraarticular complications involving the cardiovascular, pulmonary, and other organ systems. These systemic effects impose a substantial burden on patients' physical and mental well-being, as well as their socioeconomic status .The disease often affects subjects between the ages of 40 and 70; however, it can also occur at a younger age. Globally, the prevalence rate of RA is approximately 1%, with females experiencing a higher incidence . Triosephosphate isomerase (TPI) is a metabolic enzyme that regulates the flow of glycolysis and energy generation by converting dihydroxyacetone phosphate (DHAP) into D- glyceraldehyde 3-phosphate (G3P). TPI is one of the glycolytic enzymes implicated in the pathogenesis of RA.

Additionally, it has been shown to possess functions beyond glycolysis, including potential roles in the nucleus related to cancer pathogenesis and chemotherapy resistance . Some studies showed a significant correlation between elevated TPI levels and RA, with TPI serving as an independent predictor of the disease. With some findings, which include a high sensitivity of 98.5% and specificity of 100%, suggest that TPI could be a valuable biomarker for the early diagnosis and management of RA

ELIGIBILITY:
Inclusion Criteria:

- Adult patients with RA who fulfill 2010 ACR/EULAR classification criteria

Exclusion Criteria:

1. Individuals with uncontrolled chronic diseases such as hypertension , diabetes, heart disease, liver or kidney disease, other autoimmune disorders and tumors.
2. Pregnant women.
3. Rheumatologic diseases other than RA

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Adult RA patients and age- and sex-matched healthy controls will be included
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Serum Triosephosphate Isomerase (TPI) concentration (ng/mL) in Rheumatoid Arthritis (RA) patients | baseline
  This outcome assesses the quantitative difference in serum TPI concentrations, measured in nanograms per milliliter (ng/mL), between patients diagnosed with Rheumatoid Arthritis and age- and sex-matched healthy individuals.

SECONDARY OUTCOMES:
Correlation of serum TPI with Rheumatoid Arthritis disease activity markers | baseline
  This outcome assesses the association between serum TPI levels (ng/mL) and established disease activity markers in RA patients, specifically Disease Activity Score in 28 joints with ESR (DAS28-ESR)

CONTACTS AND LOCATIONS:
Overall Officials: Safaa Mahran, proff, Study Director — World Health Organization

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smolen JS, Aletaha D, Barton A, Burmester GR, Emery P, Firestein GS, Kavanaugh A, McInnes IB, Solomon DH, Strand V, Yamamoto K. Rheumatoid arthritis. Nat Rev Dis Primers. 2018 Feb 8;4:18001. doi: 10.1038/nrdp.2018.1. PMID 29417936
- [Background] Zuo J, Tang J, Lu M, Zhou Z, Li Y, Tian H, Liu E, Gao B, Liu T, Shao P. Glycolysis Rate-Limiting Enzymes: Novel Potential Regulators of Rheumatoid Arthritis Pathogenesis. Front Immunol. 2021 Nov 24;12:779787. doi: 10.3389/fimmu.2021.779787. eCollection 2021. PMID 34899740
- [Background] Escal J, Neel T, Hodin S, Boussoualim K, Amouzougan A, Coassy A, Locrelle H, Thomas T, Delavenne X, Marotte H. Proteomics analyses of human plasma reveal triosephosphate isomerase as a potential blood marker of methotrexate resistance in rheumatoid arthritis. Rheumatology (Oxford). 2024 May 2;63(5):1368-1376. doi: 10.1093/rheumatology/kead390. PMID 37527020
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Medina YF, Ruiz-Gaviria RE, Buitrago-Lopez A, Villota C. Physical articular examination in the activity of rheumatoid arthritis: a systematic review of the literature : Systematic review of the literature regarding physical examination in rheumatoid arthritis. Clin Rheumatol. 2018 Jun;37(6):1457-1464. doi: 10.1007/s10067-018-4015-4. Epub 2018 Feb 20. PMID 29464524